CLINICAL TRIAL: NCT02431832
Title: Exploration of microRNA and Metabolomics Biomarkers Predicting Drug Induced Liver Injury in Elderly People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Chung, MD, PhD, M.D., Ph.D, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DILI_Elderly
Record Dates: First submitted 2015-04-20; First posted 2015-05-01 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: Elderly
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

ARMS (1):
- Augmentin tab (Experimental)
  Interventions: Drug: Augmentin tab

INTERVENTIONS:
Drug: Augmentin tab

SUMMARY:
An open-label, one-sequence, multiple administration study for exploration of microRNA and metabolomics biomarkers to predict drug induced liver injury in healthy elderly Korean people.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, as determined by medical history, physical examination, 12-lead electrocardiogram (ECG), and clinical laboratory evaluations were eligible to participate in the study. Subjects had to be 65 to 84 years of age.

Exclusion Criteria:

* Subjects who have clinically significant disease of cardiovascular, respiratory, renal, endocrinological, hematological, gastrointestinal, neurological(central nervous system), psychiatric disorders or malignant tumor
* Subject judged not eligible for study participation by investigator

Ages: 65 Years to 84 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | up to 35 days

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seoul, South Korea